CLINICAL TRIAL: NCT06069427
Title: The Effect of Reducing Total Volume of Sprint Exercise in Sprint Interval Training Protocols on Circulating Levels of Brain-derived Neurotrophic Factor (BDNF)
Brief Title: The Effect of Reducing Total Volume of Sprint Exercise on Circulating Levels of BDNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stirling (Other)
Responsible Party: Principal Investigator, Niels Vollaard, Lecturer, University of Stirling
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14395
Record Dates: First submitted 2023-09-27; First posted 2023-10-05 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Mental Health Wellness 1
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Participants will each undergo 3 trials in a randomised order.
Masking Description: Due to the nature of the interventions (exercise), masking is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Sprint interval training (SIT) — The SIT protocol consists of 4 repeated 30-second, 'all-out' cycle sprints against a resistance equivalent to 7.5% of body mass on a stationary bicycle. The first sprint will be preceded by a 4-minute warm-up consisting of unloaded pedalling. Each sprint will be followed by 4 minutes of unloaded pedalling.
Behavioral: Reduced-exertion high-intensity interval training (REHIT — The REHIT protocol consists of 2 repeated 20-second, 'all-out' cycle sprints against a resistance equivalent to 7.5% of body mass on a stationary bicycle. The first sprint will be preceded by a 2-minute warm-up consisting of unloaded pedalling. The first sprint will be followed by 3 minutes of unloaded pedalling, and the second sprint will be followed by 4 minutes of unloaded pedalling.
Behavioral: No-exercise control (CON) — The control condition will involve seated rest for a period equivalent to the other interventions.

SUMMARY:
Regular exercise is well known to be required for good physical health, but exercise can also improve mental health. Although the effects of exercise on mental health have been shown in many studies, it remains unclear how exercise improves mental health. In recent years, the potential role of a specific protein called 'brain-derived neurotrophic factor' (BDNF) has received increasing attention. Higher levels of BDNF in the blood are associated with better cognitive performance, attention, and spatial memory. Conversely, low levels of BDNF in the blood are found in patients with depression, dementia, mild cognitive impairment, and Alzheimer's disease. BDNF can be released during exercise, with greater increases after exercise performed at higher intensities. For example, classic sprint interval training (SIT), which involves four 30-second 'all-out' cycle sprints, has been shown to lead to greater increases in BDNF compared to moderate or vigorous exercise. Although these results suggest that SIT is an effective way to increase BDNF, SIT is not generally considered feasible for patients or untrained members of the general public, because it is a very tiring type of exercise. However, other more manageable protocols have been developed, such as the 'reduced-exertion, high-intensity interval training' (REHIT) protocol, which involves two 20-second 'all-out' sprints within a 10-minute low-intensity exercise session. Although it is clear that BDNF levels increase in an intensity-dependent manner in response to exercise, the effect of exercise volume remains unknown. Exercise intensity is identical for SIT and REHIT, but if BDNF levels increase to a similar extent in response to both protocols, REHIT would constitute a more feasible intervention for use in patients and the general public. The aim of the present study is to compare the effects of REHIT vs. classic SIT on levels of BDNF in the blood. For this,15 study participants will be recruited, who will each complete a SIT session, a REHIT session, and a no-exercise control session. Levels of BDNF will be measured in blood samples taken at rest, as well as directly after exercise, 30 minutes after exercise, and 90 minutes after exercise. It will be determined whether the greater amount of sprint exercise in a SIT session will be associated with a greater increase in levels of BDNF in the blood compared to the REHIT session which consists of a lower amount of sprint exercise.

ELIGIBILITY:
Inclusion Criteria:

* Apparently health young male volunteers

Exclusion Criteria:

* Age <18 y or >40 y
* BMI > 35 kg/m2
* participation in a structured exercise training programme at any time in the preceding 6 months
* suffering from acute (e.g., common cold, Covid-19, flu, etc) or chronic disease (e.g., diabetes, heart disease, cancer, etc)
* answering 'yes' to one or more questions of a standard physical activity readiness questionnaire (PAR-Q)
* resting heart rate ≥100 bpm
* clinically significant hypertension (>140/90 mm Hg)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of BDNF | Pre-exercise, directly post-exercise, and 30 and 90 minutes post-exercise
  Plasma levels of the protein brain-derived neurotrophic factor (BDNF) will be measured pre-exercise, directly post-exercise, and 30 and 90 minutes post-exercise. The area-under-the-curve for plasma BDNF will be calculated. Differences in AUC between the 3 trails will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Vollaard, PhD, Principal Investigator — University of Stirling
Locations (1):
- University of Stirling, Stirling, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.